CLINICAL TRIAL: NCT02859662
Title: Abdominal Compartment Syndrome and Ruptured Aortic Aneurysm : Validation of a Predictive Test
Acronym: SCA-AAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: R/2015/49
Record Dates: First submitted 2016-05-09; First posted 2016-08-09 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Abdominal Compartment Syndrome
Keywords: abdominal compartment syndrome; abdominal aortic aneurysm; ruptured aneurysm
MeSH Terms: conditions — Intra-Abdominal Hypertension; Aortic Aneurysm, Abdominal; Aneurysm, Ruptured

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: ruptured aortic aneurysm — All patients with ruptured abdominal aortic aneurysm may be included in this study, whatever the surgical treatment.

SUMMARY:
It is an observational study on ruptured abdominal aortic aneurysm and abdominal compartment syndrome.

the aim of this study is to assess the qualities of a predictive score on the occurence of this syndrome after surgery of ruptured aortic aneurysm

DETAILED DESCRIPTION:
Despite improved management techniques of ruptured abdominal aortic aneurysm, especially in vascular surgery, the mortality rate has not decreased these last years.

The abdominal compartment syndrome (ACS) has been clearly identified as one of the main etiologies of mortality after ruptured aortic aneurysm. The mortality grow up with ACS in this population.

So, the investigators want to screen abdominal compartment syndrome in the operative room.

It is an observational study on ruptured abdominal aortic aneurysm and abdominal compartment syndrome.

the aim of this study is to assess the qualities of a predictive score on the occurence of this syndrome after surgery of ruptured aortic aneurysm

Later the aim of a future study will be to screen ACS and manage patient as soon as possible to avoid it.

ELIGIBILITY:
Inclusion Criteria:

* over 18
* to be hospitalized in participating hospitals
* ruptured aneurysm confirmed and operated

Exclusion Criteria:

* pregnancy
* patients with bladder tumor or bladder surgery or trauma bladder can distort bladder pressure measurement
* cystectomy
* patients died before arrival in the operating room
* patients died during surgery or within one hour of the initial surgical procedure
* patient whose abdominal closure at the end of the procedure is impossible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with ruptured abdominal aortic aneurysm may be included in the study, whatever the surgical technique used.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
a predictive score on the appearance of an abdominal compartment syndrome after a surgical treatment of a ruptured abdominal aortic aneurysm | 30 days
  score with criteria

SECONDARY OUTCOMES:
30 days mortality rate | 30 days
  Mortality
the duration of hospitalisation (intensive care unit stay and total hospital stay) | 30 days
  Duration in day of hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Simon Rinckenbach, MD PhD, Principal Investigator — CHRU Besancon
Locations (10):
- France (10):
  - CHU, Bordeaux
  - CHU, Clermont-Ferrand
  - CH, Colmar
  - CHU, Dijon
  - CHU, Lyon
  - CH, Mulhouse
  - CHU, Nancy
  - CHU, Nantes
  - CHU, Rennes
  - CHU Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leclerc B, Salomon Du Mont L, Parmentier AL, Besch G, Rinckenbach S. Abdominal compartment syndrome and ruptured aortic aneurysm: Validation of a predictive test (SCA-AAR). Medicine (Baltimore). 2018 Jun;97(25):e11066. doi: 10.1097/MD.0000000000011066. PMID 29923999